CLINICAL TRIAL: NCT05653050
Title: An Open-label, Multi-centre, Randomised, Two-period, Crossover Study to Assess the Efficacy, Safety and Utility of Closed-loop Glucose Control Compared to Standard Insulin Pump Therapy Combined with Continuous Glucose Monitoring in Adolescents with Type 1 Diabetes
Brief Title: Closing the Loop in People with Type 1 Diabetes
Acronym: CLEAR Phase 2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cambridge (Other)
Collaborators: Manchester University NHS Foundation Trust (Other Government); Barts & The London NHS Trust (Other); Norfolk and Norwich University Hospitals NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Dr Roman Hovorka, Professor, University of Cambridge
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CLEAR Phase 2
Record Dates: First submitted 2022-11-09; First posted 2022-12-16 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Continuous Glucose Monitoring

STUDY DESIGN:
Intervention Model Description: An open-label, multi-centre, randomised, two-period, crossover study comparing fully closed-loop glucose control to standard insulin pump therapy combined with continuous glucose monitoring
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Fully closed-loop system with age-approved ultra-rapid insulin (Experimental): The fully closed-loop system (CamAPS HX) will consist of:
  * Mylife YpsoPump insulin pump (Ypsomed, Burgdorf, Switzerland).
  * Freestyle Libre 3 real-time CGM sensor (Abbott, Diabetes Care, CA, USA)
  * Android smartphone hosting CamAPS HX App with the Cambridge model predictive control algorithm.
  * Cloud upload system to review CGM/insulin data.
  Participants will use ultra-rapid insulin aspart in the closed-loop system.
  Interventions: Device: CamAPS HX
- Standard insulin pump therapy with CGM (Active Comparator): Participants will use their own insulin pump and usual insulin throughout this study period.
  The CGM will be the Freestyle Libre 3 real-time CGM sensor (Abbott, Diabetes Care, CA, USA).
  Interventions: Device: Standard insulin pump therapy with CGM

INTERVENTIONS:
Device: CamAPS HX — Fully automated closed-loop system (CamAPS HX) with ultra-rapid insulin aspart.
  Arms: Fully closed-loop system with age-approved ultra-rapid insulin
Device: Standard insulin pump therapy with CGM — Participants usual insulin pump therapy with Freestyle Libre 3 CGM
  Arms: Standard insulin pump therapy with CGM

SUMMARY:
The main objective of this study is to determine whether home use of fully closed-loop glucose control applying age-approved ultra-rapid insulin (Phase 2) is superior to standard insulin pump therapy with continuous glucose monitoring (CGM) in adolescents with type 1 diabetes on insulin pump therapy with sub-optimal glycaemic control (HbA1c ≥ 7.5% [Phase 2]).

This is an open-label, multi-centre, randomised, crossover design study, involving a run-in period followed by two study periods during which glucose levels will be controlled either by an automated closed-loop system using age-approved ultra-rapid insulin or by participants' usual insulin pump therapy with continuous glucose monitoring in random order. A total of up to 30 adolescents (aiming for 24 completed participants) with T1D on insulin pump therapy will be recruited through diabetes clinics and other established methods.

Participants will receive appropriate training in the safe use of the closed-loop devices. Participants will have access to the study team during the home study phase with 24/7 telephone support.

The primary outcome is time spent in target range between 3.9 and 10.0 mmol/L as recorded by CGM over the 8 week period. Secondary outcomes are HbA1c, time spent with glucose levels above and below target as recorded by CGM, and other CGM-based metrics in addition to insulin requirements. Safety evaluation comprises severe hypoglycaemic episodes, diabetic ketoacidosis (DKA) events and other adverse and serious adverse events.

DETAILED DESCRIPTION:
Purpose of clinical trial:

To determine whether home use of fully closed-loop applying age-approved ultra-rapid insulin is superior to insulin pump therapy with continuous glucose monitoring (CGM).

Study objectives:

The study objective is to compare home use of fully closed-loop glucose control applying ultra-rapid Lispro insulin (Phase 1) or age-approved ultra-rapid insulin (Phase 2) with standard insulin pump therapy with CGM.

1. EFFICACY: The objective is to assess the efficacy of fully closed-loop glucose control applying ultra-rapid Lispro insulin (Phase 1) or age-approved ultra-rapid insulin (Phase 2) in maintaining CGM glucose levels within the target range from 3.9 to 10.0 mmol/l, as compared to standard insulin pump therapy combined with CGM.
2. SAFETY: The objective is to evaluate the safety of fully closed-loop glucose control in terms of episodes of severe hypoglycaemia, hyperglycaemia and other adverse events and adverse device effects.
3. UTILITY: The objective is to determine the percentage of time when closed-loop was operational, and usability and acceptance of the closed-loop system.

Participating clinical centres:

1. Addenbrooke's Hospital, Cambridge University Hospitals NHS Foundation Trust, Cambridge
2. Diabetes, Endocrine & Metabolism Centre, Manchester Royal Infirmary, Manchester University NHS Foundation Trust, Manchester
3. Alder Hey Children's NHS Foundation Trust, Liverpool.
4. The Royal London Children's Hospital of Whitechapel Road, Barts Health NHS Trust, London

Sample Size:

24 adolescents completing the study. Up to 30 for phase 2 will be recruited to allow for dropouts.

Maximum duration of study for a participant:

20 weeks (5 months)

Recruitment:

The participants will be recruited through the young adult and paediatric diabetes outpatient clinics or other established methods.

Consent:

Participants and/or parents/guardians will be asked to provide written informed consent/assent.

Baseline Assessment:

Eligible participants will undergo a baseline evaluation including a blood sample for the measurement of HbA1c, renal, thyroid functions and coeliac antibody screen (if not done in the previous 6 months). Urine pregnancy test will be done in females of child bearing age. Human factor questionnaires will be administered.

Run-in Period:

During the 2-3 week run-in period, participants will use their own insulin pump and wear a masked CGM system. At the end of the run-in period, for compliance, at least 10 days of CGM data need to be recorded. CGM data during the run-in period will be used to assess baseline glucose control before the start of the first home study phase.

Randomisation:

Eligible participants will be randomised using randomisation software to the use of closed-loop glucose control or to standard pump therapy with CGM. There will be no washout period between the two intervention periods.

1. Automated closed-loop:

   Training on the use of closed-loop will be provided by the research team during a 2 to 3 hour session in an outpatient setting (clinical research facility) or may be done remotely/at home. Competency on the use of study insulin pump, study CGM and closed-loop system will be evaluated using a competency assessment tool developed by the research team. Further training may be delivered as required. Participants will be advised to use the closed-loop system with age-approved ultra-rapid insulin for the next 8 weeks.
2. Conventional insulin pump therapy with CGM:

Participants will use their own insulin pump and study CGM. Training on the use of real-time CGM and how to interpret real-time will be provided. Participants will use standard insulin pump therapy, with their usual insulin, and real-time CGM for the next 8 weeks.

Cross-over Assessment:

At the end of the first intervention period, a blood sample for the measurement of HbA1c will be taken and human factor questionnaires will be administered.

End of study assessments:

A blood sample will be taken for measurement of HbA1c and human factor questionnaires will be administered. Study devices will be returned and participants will resume usual care.

Procedures for safety monitoring during trial:

Standard operating procedures for monitoring and reporting of all adverse events and adverse device events will be in place, including serious adverse events (SAE), serious adverse device effects (SADE) and specific adverse events (AE) such as severe hypoglycaemia.

A data monitoring and ethics committee (DMEC) will be informed of all serious adverse events and any unanticipated adverse device/method effects that occur during the study and will review compiled adverse event data at periodic intervals.

Criteria for withdrawal of patients on safety grounds:

A participant may terminate participation in the study at any time without necessarily giving a reason and without any personal disadvantage. An investigator can stop the participation of a subject after consideration of the benefit/risk ratio. Possible reasons are:

* Serious adverse events
* Significant protocol violation or non-compliance
* Failure to satisfy competency assessment
* Decision by the investigator, or the sponsor, that termination is in the participant's best medical interest
* Pregnancy, planned pregnancy, or breast feeding
* Allergic reaction to insulin
* Technical grounds (e.g. participant relocates)

ELIGIBILITY:
Inclusion Criteria:

* The participant has type 1 diabetes as defined by WHO for at least 1 year
* The participant is aged 13 to 19 years (inclusive) (Phase 2)
* The participant will have been on an insulin pump for at least 3 months with good knowledge of insulin self-adjustment
* The participant is treated with one of the rapid acting or ultra-rapid acting insulin analogues (Insulin Aspart, faster acting insulin Aspart, Insulin Lispro, ultra-rapid Lispro insulin or Insulin Glulisine) 6. HbA1c ≥7.5% (58mmol/mol) based on analysis from local laboratory 7. The participant is willing to wear closed-loop devices 8. The participant is willing to follow study specific instructions 9. Female participants of child bearing age must have a negative urine-HCG pregnancy test at screening and should be using effective contraception if sexually active.

Exclusion Criteria:

1. Any physical or psychological disease or condition likely to interfere with the normal conduct of the study and interpretation of the study results
2. Known or suspected allergy against insulin
3. Total daily insulin dose more than or equal to 2 IU/kg/day
4. Use of a closed-loop system within the past 30 days
5. Participant is pregnant or breast feeding or planning pregnancy within next 12 months
6. Severe visual impairment
7. Severe hearing impairment
8. Lack of reliable telephone facility for contact
9. Participant not proficient in English

Ages: 13 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 26 (Actual)
Dates: Start 2023-02-20 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-10-15 (Actual)

PRIMARY OUTCOMES:
Time in target glucose range | 8-week home use
  Time spent in the target glucose range from 3.9 to 10.0 mmol/l (70 to 180mg/dl) based on continuous glucose monitoring (CGM)

SECONDARY OUTCOMES:
Time spent above the target glucose range | 8-week home use
  Time spent above target glucose (10.0 mmol/l) (180 mg/dl) based on CGM
Time spent below the target glucose range | 8-week home use
  Time spent below target glucose (3.9 mmol/l) (70 mg/dl) based on CGM
Mean glucose | 8-week home use
  Average of sensor glucose levels
Standard deviation and coefficient of variation of glucose | 8-week home use
  Standard deviation and coefficient of variation of CGM glucose levels
Time spent in hypoglycaemia | 8-week home use
  Time with glucose levels < 3.5 mmol/l (63mg/dl), < 3.0 mmol/l (54mg/dl), and <2.8 mmol/l (50mg/dl) based on CGM
Time spent in hyperglycaemia | 8-week home use
  Time with glucose levels in the significant hyperglycaemia (glucose levels > 20.0 mmol/l) (360mg/dl)
HbA1c | After 8-week home use
  Glycated haemoglobin measured at the end of the treatment period(360mg/dl)
Total, basal, and bolus insulin dose | 8-week home use
  Total, basal, and bolus insulin dose

OTHER OUTCOMES:
Safety evaluation | 8-week home use
  The number of episodes of severe hypoglycaemia events
Safety evaluation | 8-week home use
  The number of episodes of DKA events
Safety evaluation | 8-week home use
  The number of episodes of significant ketonemia (> 3.0mmol/l) events
Safety evaluation | 8-week home use
  The number and nature of any other adverse events
Safety evaluation | 8-week home use
  The number of SADEs
Utility evaluation | 8-week home use
  Frequency and duration of use of the closed-loop system at home The number of episodes of hypoglycaemia, DKA and / or significant ketonemia (> 3.0mmol/l) as well as nature and severity of any other adverse events including SADEs and SAEs.
Human Factor assessment | After 8-week home use
  Expectations, attitudes and responses to the closed-loop system will be assessed using the INSPIRE questionnaire.
Human Factor assessment | After 8-week home use
  Diabetes distress will be assessed using the PAID-Teen questionnaire.
Human Factor assessment | After 8-week home use
  Hypoglycemia fear will be assessed using the Hypoglycemia Fear Survey (HFS II) Child version

CONTACTS AND LOCATIONS:
Locations (4):
- United Kingdom (4):
  - Addenbrooke's Hospital, Cambridge
  - Barts Health NHS Trust, London
  - Manchester Royal Infirmary, Manchester
  - Norfolk and Norwich University Hospitals NHS Foundation Trust, Norwich

IPD SHARING:
Plan to Share IPD: Yes
Study protocol, statistical analysis plan and fully anonymised individual participant data that underlie the results reported in the manuscript will be available 6 months following publication and ending 36 months following manuscript publication to investigators whose proposed use of the data has been approved by an independent review committee identified for this purpose, to achieve aims in the approved proposal. Proposals should be directed to rh347@cam.ac.uk and may be submitted up to 36 months following article publication. To gain access, data requestors will need to sign a data access agreement.
  Fully anonymised data may be shared with third parties (EU or non-EU based) for the purposes of advancing management and treatment of diabetes.
Supporting Information: Study Protocol, SAP
Time Frame: Study protocol, statistical analysis plan and fully anonymised individual participant data that underlie the results reported in the manuscript will be available 6 months following publication and ending 36 months following manuscript publication to investigators whose proposed use of the data has been approved by an independent review committee identified for this purpose, to achieve aims in the approved proposal. Proposals should be directed to rh347@cam.ac.uk and may be submitted up to 36 months following article publication.
Access Criteria: Study protocol, statistical analysis plan and fully anonymised individual participant data that underlie the results reported in the manuscript will be available 6 months following publication and ending 36 months following manuscript publication to investigators whose proposed use of the data has been approved by an independent review committee identified for this purpose, to achieve aims in the approved proposal. Proposals should be directed to rh347@cam.ac.uk and may be submitted up to 36 months following article publication.

REFERENCES:
- [Derived] Kadiyala N, Allen J, Lakshman R, Boughton CK, Wilinska ME, Thankamony A, Hartnell S, Thabit H, Willemsen RH, Shah P, Ware J, Hovorka R. Lived experience of fully closed-loop insulin delivery in adolescents with type 1 diabetes and HbA1c above target. Diabetes Res Clin Pract. 2025 Dec 30;232:113078. doi: 10.1016/j.diabres.2025.113078. Online ahead of print. PMID 41478508